CLINICAL TRIAL: NCT00002693
Title: PHASE I STUDY OF CONTINUOUS INFUSION CARBOPLATIN AND TOPOTECAN IN THE TREATMENT OF RELAPSED ACUTE LEUKEMIA AND BLAST CRISIS CHRONIC MYELOGENOUS LEUKEMIA
Brief Title: Combination Chemotherapy in Treating Patients With Chronic Myelogenous Leukemia or Recurrent Acute Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scott Harold Kaufmann, M.D. Ph.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000064447; U01CA069912 (NIH); P30CA015083 (NIH); 958101 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-04-11 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Leukemia; Neutropenia
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; neutropenia
MeSH Terms: conditions — Leukemia; Neutropenia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Blast Crisis | interventions — Filgrastim; Carboplatin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy with carboplatin and topotecan in treating patients with chronic myelogenous leukemia or recurrent acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the maximum tolerated dose of carboplatin plus topotecan given as a 5-day continuous infusion in patients with recurrent acute lymphocytic or myeloid leukemia or accelerated or blastic phase chronic myelogenous leukemia.
* Assess the toxicity of this regimen in these patients.
* Gather preliminary information on the activity of this regimen in these patients.
* Examine the pharmacokinetics of topotecan when administered concurrently with carboplatin.

OUTLINE: This is a dose escalation study of topotecan. Patients are stratified according to prior bone marrow transplant (BMT) (yes vs no).

* Induction: Patients receive carboplatin and topotecan IV 3 times a day on days 1-5. Patients may also receive filgrastim (G-CSF) beginning on day 7 or 14. Retreatment is based on results of marrow exam on day 10-14. Patients with less than 5% blasts undergo a second marrow exam upon blood count recovery or on day 26-30, whichever is earlier. Patients with at least 5% blasts after day 21 receive one more course, in the absence of unacceptable toxicity and at the discretion of the investigator. Patients with no greater than 5% blasts begin G-CSF if blood counts are not recovered, then proceed to consolidation.

Cohorts of 1-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of up to 6 patients experience dose limiting toxicity. Patients with prior BMT will not be entered at any level until 3-6 patients with no prior BMT tolerate that level.

* Consolidation (begins around day 42 of last Induction course): Patients with ALL/AML in complete remission (CR) or CML in chronic phase receive 2 additional courses (same doses) 6-8 weeks apart.

Patients experiencing a relapse after CR lasting at least 6 months may receive additional treatment.

PROJECTED ACCRUAL: A total of 15-20 patients without and 2-20 patients with prior bone marrow transfer will be accrued for this study over 2-2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute lymphocytic or myeloid leukemia (ALL or AML) in 1 of the following categories:

  * Failed to achieve a complete response (CR) with initial induction regimen
  * First relapse within 1 year of initial CR
  * Failed re-induction therapy at first relapse
  * Second relapse after no more than 2 different induction regimens
  * Relapse defined as more than 10% blasts in marrow or circulating blasts in peripheral blood and either:

    * Symptoms of recurrence (e.g., B symptoms)
    * Evidence of impending marrow failure (i.e., cytopenias) OR
* Chronic myelogenous leukemia in accelerated or blastic phase after no more than 1 prior induction regimen
* No HLA-identical sibling marrow donor or patient ineligible for allogeneic marrow transplantation
* No clinical symptoms of CNS leukemia

  * Patients with history of CNS leukemia must have pretreatment lumbar puncture demonstrating absence of active CNS disease
* No active CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 4 weeks

Hematologic:

* Not applicable

Hepatic:

* Bilirubin less than 2 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No congestive heart failure
* No poorly controlled arrhythmia
* No myocardial infarction within the past 3 months

Other:

* No active infection
* No other serious medical condition that would prevent compliance
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 24 hours since prior hydroxyurea for impending leukostasis
* No concurrent hydroxyurea glucocorticoids
* Recovered from prior chemotherapy

Endocrine therapy:

* At least 24 hours since prior glucocorticoids for impending leukostasis
* At least 7 days since prior amphotericin or aminoglycosides
* No concurrent glucocorticoids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No concurrent aminoglycoside antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H. Kaufmann, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Kaufmann S, Letendre L, Litzow M, et al.: Phase I study of continuous infusion (CI) topotecan (TPT) and carboplatin (CBDCA) for relapsed or refractory acute leukemia. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A107, 1998.